CLINICAL TRIAL: NCT04096170
Title: Improving Pain Control in Paraesophageal Hernia Repair: Intravenous Lidocaine Versus Placebo
Acronym: PEH
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00081332; 06-18-03 (Other: Atrium); Pro00027862 (Other: Atrium)
Record Dates: First submitted 2019-09-18; First posted 2019-09-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Hernia, Paraesophageal
MeSH Terms: conditions — Hernia, Hiatal | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV Lidocaine (Experimental): 100 mg Lidocaine bolus on induction, then an infusion of 1.5 mg/kg/hr to begin prior to incision, run throughout the operation and continues into PACU for 1 hour OR until one 2gm/250mL D5W bag has been infused, whichever occurs first. The Patient will be monitored by nursing staff with the aid of continuous cardiac monitoring in the PACU for at least 30 minutes after the discontinuation of the lidocaine drip.
  Interventions: Drug: IV lidocaine
- Placebo (Placebo Comparator): Patients will receive D5W solution at the same volume and rate as the IV lidocaine.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IV lidocaine — Patients randomized to the IV lidocaine group will receive a 100 mg lidocaine bolus on induction then an infusion of 1.5 mg/kg/hr prior to incision. This infusion will continue throughout operation and into the PACU for 1 hour OR until the 2gm/250 mL D5W bag has been infused, whichever occurs first.
  Arms: IV Lidocaine
Drug: Placebo — o Patients randomized to the placebo group will receive D5W solution (as this is the carrier for lidocaine) at the same volume and rate as the IV lidocaine.
  Arms: Placebo

SUMMARY:
We aim to study the impact of perioperative IV lidocaine on postoperative pain control in patients undergoing paraesophageal hernia repair. This is in the context of an established ERAS protocol. We wish to study the effect of IV Lidocaine on postoperative short and long-term outcomes, including patients' length of stay postoperative mortality, morbidity, and quality of life. We will compare this to our standard pain management.

DETAILED DESCRIPTION:
Patients will be prospectively enrolled from Carolinas Hernia Center's outpatient clinic. All paraesophageal hernia patients, age 18 and older, undergoing PEH repair at CHS will be included. We will conduct a two-arm prospective randomized study, IV Lidocaine versus placebo, to study the reduction of narcotics, return to bowel function and length of stay. Both arms will receive standard multimodal pain control in the operative and postoperative period. There will be two arms: 1. IV Lidocaine 2. Placebo. Subject participation will last approximately 6 months for this study. Lidocaine will be used as a perioperative adjunct. At the conclusion of the study, chart review will be performed to evaluate if Lidocaine infusion limited narcotic need, or effected Visual Analog Scale (VAS) values. VAS is the standard nursing method of documenting pain using pain scores. The nurses ask the patient to rate pain from 0 (no pain) to 10 (excruciating pain). LOS is a secondary endpoint of the study, as subjects in the lidocaine arm are hypothesized to have improved pain control and require lower narcotic dosing, potentially leading to earlier discharge. We will evaluate patient demographics, preoperative lab values, intraoperative and perioperative variables, as well as postoperative outcomes and pain reported by VAS. Postoperative data to be reviewed will also include total opioid analgesia administered, time from surgery to a clear liquid diet, time from surgery to a post-fundoplication diet, time to return of bowel function, length of stay, pain/VAS scores at 6 hours postoperatively, pain/VAS scores on each post-operative day until discharge, pain/VAS scores at 2 and 4 weeks, and pain/VAS scores at 6 months, infectious complications (urinary tract infections as well as surgical site infections, deep organ space infections, pneumonia), and non-infectious complications (stroke, myocardial infarction, respiratory failure, post-op bleeding, unplanned return to the OR, acute renal failure, death, etc.). When results of the study are published, the subject's identity will remain confidential. Data will be analyzed using standard statistical methods; all patient-identifying information will be removed prior to analysis. Descriptive statistics including means and standard deviations, medians and interquartile range, or counts and percentages, will be used to describe the study population on all variables. For continuous variables comparisons will be made between groups using t-tests and Wilcoxon Rank Sum test. For categorical variables, Chi-Square test and Kruskal-Wallis tests will be used for comparisons between groups. Multivariate regression will be performed as needed to control for potential confounding factors such as age, gender and type of procedure. A p-value of <0.05 will be used for all significance determinations. The SAS® system version 9.4 (Cary, NC) or similar program will be used to complete all statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18+ years of age
* American Association of Anesthesiologists (ASA) scores of I-III
* Undergoing elective laparoscopic paraesophageal hernia repair including robotic assisted laparoscopic cases.
* All paraesophageal hernia patients seen in clinic who meet inclusion criteria will be given the option to enroll.
* Cases converted to open laparotomy or hand-assisted laparoscopy will be included for intention to treat analysis.
* Patients who have complications of Clavien-Dindo class 3 or greater will be included in calculations of complication rates. However, they will not be included in calculations of postoperative morphine equivalents, as repeat intervention will confound the normal course of postoperative pain control.

Exclusion Criteria:

* Patients with end stage renal disease
* Patients with allergies to lidocaine and other amide local anesthetics.
* Patients with contraindications to sodium channel blockers.
* Patients with psychomotor retardation
* Patients with body mass index >40 mg/kg2.
* Patients receiving opioid pain medication in the previous week or taking daily medication for chronic pain
* Patients with a seizure disorder
* Patients with cardiac intraventricular conduction delays, congestive heart failure, first and second-degree heart conduction blocks.
* Patients undergoing planned concomitant procedures other than PEH repair
* Patients that are classified as ASA 4 or 5 during pre-operative anesthesia visit (if needed) will be excluded. Documentation from the pre-op visit will be reviewed by the research team prior to the surgery date.
* Exclusion from all or portions will be at the discretion of the attending surgeon and anesthesiologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-06-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Post-Op Morphine Equivalents | Post-operation up to 6 months
  Post-operative consumption of morphine equivalents
VAS Pain Score | post-op to 6 months
  VAS is the standard nursing method of documenting pain using pain scores. The nurses ask the patient to rate pain from 0 (no pain) to 10 (excruciating pain).
Length of Stay | up to 6 months
  Length of stay post op
Return of bowel function | up to 6 months
  We will track when each patient passes first bowel movement expressed as hours since operation
Day to toleration of diet | up to 6 months
  When the patient tolerates a normal diet

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Colavita, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health - Carolinas Medical Center, Charlotte, North Carolina, United States